CLINICAL TRIAL: NCT05126173
Title: A Clinical Validation Study to Demonstrate the Effectiveness of an Artificial Intelligence Algorithm (DERM) to Identify Skin Cancer in Patients Undergoing a Skin Biopsy
Brief Title: DERM US and EU Validation Study
Status: Completed | Type: Observational
Sponsor: Skin Analytics Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: DERM-006
Record Dates: First submitted 2021-10-18; First posted 2021-11-18 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Malignant Skin Melanoma T0; Basal Cell Carcinoma; Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Deep Ensemble for the Recognition of Malignancy (DERM) — An AI-based diagnosis support tool

SUMMARY:
This study aims establish the effectiveness of Image Analysing Algorithm (DERM) to identify melanoma, Squamous Cell Carcinoma (SCC) and Basal Cell Carcinoma (BCC) when used to analyse dermoscopic images of skin lesions within the US and European population.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study,
* Male or Female, aged 18 years or above,
* Have at least one suitable skin lesion that will be biopsied due to a suspicion of skin cancer,

To be suitable for inclusion, a skin lesion must NOT have ANY of the following limitations:

located on an anatomical site of different skin structure: palms of hands or soles of feet (acral lesion), mucosal surfaces (lips and eyes) or under nail (ungal lesion), a diameter greater than the diameter of the dermoscopic lenses, located on an anatomical site unsuitable for photographing, including on surface of genitals and hair-bearing areas, has been previously biopsied, excised, treated or otherwise traumatised, located in an area of visible scarring or tattooing.

- In the Investigator's opinion, able and willing to comply with all study requirements.

Exclusion Criteria:

* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients attending a dermatology clinic with at least one skin lesion that will be biopsied due to a suspicion of skin cancer will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 1111 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity of DERM to detect "Malignant conditions" | Through study completion, on average of 1 day
  Sensitivity of DERM to detect Melanoma, SCC and BCC combined
Specificity of DERM to detect Malignant conditions. | Through study completion, on average of 1 day
  Specificity of DERM to detect Melanoma, SCC and BCC combined

SECONDARY OUTCOMES:
Sensitivity of DERM to detect Melanoma | Through study completion, on average of 1 day
  Sensitivity of DERM to detect Melanoma
Specificity of DERM to detect Melanoma | Through study completion, on average of 1 day
  Specificity of DERM to detect Melanoma
Sensitivity of DERM to detect Squamous Cell Carcinoma | Through study completion, on average of 1 day
  Sensitivity of DERM to correctly classify SCC
Specificity of DERM to detect Squamous Cell Carcinoma | Through study completion, on average of 1 day
  Specificity of DERM to correctly classify SCC
Sensitivity of DERM to detect Basal Cell Carcinoma | Through study completion, on average of 1 day
  Sensitivity of DERM to correctly classify BCC
Specificity of DERM to detect Basal Cell Carcinoma | Through study completion, on average of 1 day
  Specificity of DERM to correctly classify BCC
Accuracy of mole/not mole algorithm | Through study completion, on average of 1 day
  Accuracy of mole/not mole algorithm

OTHER OUTCOMES:
Diagnostic accuracy measures | Through study completion, on average of 1 day
  AUROC, sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) etc. of DERM to detect melanoma, SCC, BCC, premalignant, and benign conditions grouped and individually
Probability that the most probable lesion label DERM returns matches the lesion diagnosis | Through study completion, on average of 1 day
  Probability that the alternative classification label DERM that returns, matches the lesion diagnosis
The impact of patient characteristics on the diagnostic accuracy of DERM | Through study completion, on average of 1 day
  Such as sex, age, and Fitzpatrick skin type
The impact of lesions characteristic on the diagnostic accuracy of DERM | Through study completion, on average of 1 day
  Such as location, size, growth, stage and sub-type
AUROC of DERM to identify malignant conditions for each individual camera / lens type | Through study completion, on average of 1 day
  AUROC of DERM to identify malignant conditions for each individual camera / lens type
Concordance of DERM results by each individual camera / lens type | Through study completion, on average of 1 day
  Concordance of DERM results by each individual camera / lens type
Strength of association between correct classification and acceptance/rejection status of images | Through study completion, on average of 1 day
  Strength of association between correct classification and acceptance/rejection status of images
AUROC of DERM when macro images are used both to train the algorithm and as test images | Through study completion, on average of 1 day
  AUROC of DERM when macro images are used both to train the algorithm and as test images
Correlation between clinician assessment of likelihood of skin cancer with histopathology diagnosis | Through study completion, on average of 1 day
  Correlation between clinician assessment of likelihood of skin cancer with histopathology diagnosis
Percentage of images taken that are rejected by the IQ check (MoleNotMole + Image Quality), where a second image is successfully taken | Through study completion, on average of 1 day
  Percentage of images taken that are rejected by the IQ check (MoleNotMole + Image Quality), where a second image is successfully taken

CONTACTS AND LOCATIONS:
Locations (16):
- United States (10):
  - Stanford university, Redwood City, California
  - Vista Health Research, LLC, Miami, Florida
  - Dorisca Research Consulting, LLC, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - ALLCUTIS Research, LLC, Beverly, Massachusetts
  - Allcutis Research, Methuen, Massachusetts
  - Universal Dermatology, PLLC, Fairport, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Alpesh D. Desai, DO, PLLC, a Houston company institution, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Italy (6):
  - Universitaria Di Bologna, Bologna
  - Dermatology University of Florence, Florence
  - Università degli Studi di Modena e Reggio Emilia, Modena
  - University of Campania, Napoli
  - Università del Piemonte Orientale, Novara
  - UOSD Dermatology Oncology, Roma